CLINICAL TRIAL: NCT00912457
Title: Donepezil Treatment for Sleep Apnea Patients: A Double Blind Placebo-Controlled Study
Brief Title: Donepezil Treatment for Sleep Apnea Patients
Acronym: doneapnea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associacao Fundo de Incentivo a Psicofarmcologia (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Walter Andre dos Santos Moraes, AFIP
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP0043/07
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: sleep apnea; donepezil; pharmacological; cholinergic
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil (Experimental): Donepezil-treated sleep apnea patients
  Interventions: Drug: donepezil
- Placebo (Placebo Comparator): Placebo-treated sleep apnea patients
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: donepezil — donepezil 5 mg/day for 14 days followed by donepezil 10 mg/day for 14 days
  Other Names: Eranz, Aricept
  Arms: Donepezil
Drug: placebo — placebo 1 p/day for 28 days
  Other Names: Non-active substance
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of the anticholinesterase drug donepezil on sleep apnea patients. Sleep structure and respiratory parameters will be analyzed by polysomnography.

DETAILED DESCRIPTION:
Cholinergic activity also influences the upper airway opening via central and peripheral mechanisms. Decreased thalamic pontine cholinergic projections may affect respiratory drive leading to both central and obstructive apnea at least in certain degenerative conditions.In contrast to the prolific literature on physical and surgical treatments for sleep apnea there is a dearth of effective pharmacological approaches.Most drugs previously tested for this purpose acted upon monoaminergic and adenosinergic systems and showed unsuccessful or ambiguous results.A previous study showed that donepezil treatment improved apnea-hypopnea index and oxygen saturation in patients with Alzheimer's disease. Treatment also increased REM sleep duration and reduced ADAS-cog scores.Based on these facts we hypothesize that donepezil treatment may be beneficial for sleep apnea patients.

Intervention: Patients will be administered donepezil or placebo. The study has a randomized, double-blind placebo-controlled design. Complete polysomnography will be performed at baseline, after 28 days of drug or placebo treatment, after 15 days drug or placebo washout and after 28 days of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of obstructive sleep apnea according to American Academy of Sleep Medicine criteria

Exclusion Criteria:

* body mass index > 40
* use of psychoactive drugs
* presence of neurological, cardiological and pulmonary diseases

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Polysomnography parameters: respiratory parameters, sleep structure | baseline, 28 days, 15 days, 28 days

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | baseline, 28 days, 15 days, 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Walter Moraes, MD PhD, Principal Investigator — Associacao Fundo de Incentivo a Psicofarmcologia; Lucia Sukys-Claudino, MD, Study Director — AFIP / UNIFESP; Dalva Poyares, MD, PhD, Study Chair — AFIP/ UNIFESP; Sergio Tufik, MD, PhD, Study Chair — AFIP/ UNIFESP
Locations (1):
- Instituto do Sono / Associacao Fundo de Incentivo a Psicofarmacologia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sukys-Claudino L, Moraes W, Guilleminault C, Tufik S, Poyares D. Beneficial effect of donepezil on obstructive sleep apnea: a double-blind, placebo-controlled clinical trial. Sleep Med. 2012 Mar;13(3):290-6. doi: 10.1016/j.sleep.2011.09.014. Epub 2012 Jan 26. PMID 22281004